CLINICAL TRIAL: NCT04325555
Title: Pre-exposure Prophylaxis: A Miracle Drug or a Moral Hazard
Status: Completed | Type: Observational
Sponsor: New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 097-2018
Record Dates: First submitted 2020-02-29; First posted 2020-03-27 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Syphilis; Chlamydia; Gonorrhea; Sexually Transmitted Diseases
MeSH Terms: conditions — Syphilis; Chlamydia Infections; Gonorrhea; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Respondents on PrEP: On PrEP status will be operationalized in multiple ways, and sensitivity analyses will be conducted using multiple definitions as a result of the self-reported nature of the study.
  1. Respondents "on PrEP" are respondents who reported that they are currently on PrEP
  2. Respondents "on PrEP" are respondents who reported to have ever been on PrEP
  3. When respondents are used as their own controls, years on PrEP will be those in which they reported to have been on PrEP for at lest 6 months, and PrEP initiation will be the first such year
  A comparison group will be constructed by matching on a variety of characteristics, when this method is applied. Most importantly, age, and STD testing frequency among others, which influence the likelihood of being on PrEP and via that avenue sexual practices, as well as the likelihood of detecting STDs (i.e., ascertainment bias). In other models adjustments will be made for these factors.
  Interventions: Drug: PrEP

INTERVENTIONS:
Drug: PrEP — The investigators measure self-reported PrEP status as exposure, i.e., PrEP status is not confirmed via matched medical records or any other type of information directly collected form subjects.

SUMMARY:
The investigators study the behavioral consequences of Pre-exposure Prophylaxis or PrEP on sexual health behaviors, sexual health outcomes, and partner selection preferences. The study collects observational, self-reported data on PrEP status, PrEP taking-history, PrEP adherence over the last 30 days, STD diagnosis history dating back to January 2015 up to December 2019, sexual health behaviors (e.g., positioning, number of lifetime/recent partners, condom adherence etc.), and various demographic characteristics. The survey finishes with a conjoint experiment which asks respondents to select between two potential partners, and follow-up question about each profiles. Potential partners' characteristics include recreational drug use and condom adherence. Recruitment is conducted via running an ad on Facebook in New York, London, Toronto and Sydney for comparative purposes, as these metro areas have varying levels of PrEP use and accessibility.

DETAILED DESCRIPTION:
See statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above
* living in the London, New York, Toronto or Sydney metro area
* self-reported sex at birth is male
* reported ever having sex with a male

Exclusion Criteria:

* not meeting the inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The survey is being distributed via Facebook ads, which are geographically targeted in the above-mentioned metro areas, with filters set up to target specifically males who are likely to be men who have sex with men (MSM). This latter is achieved by setting up a long list of sites that have been liked or followed, which map onto sexual orientation. The survey is incentivized with an Amazon gift card to be given to a randomly selected participant in each of the geographic areas after completion. Those who click on the ad are directed to the survey. They first receive questions that gauges their eligibility, and in case they are not eligible, they are screened out of the survey, and are not eligible to enroll in the raffle for the gift card, which is only available for those who finished the sutdy.
Sampling Method: Non-Probability Sample
Enrollment: 2647 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Syphilis diagnosis | All diagnosis data is collected in a time-stamped fashion between January 2015 and December 2019; diagnosis is reported within the year, but not in a specific month/day
  Self-reported diagnosis of syphilis
Chlamydia diagnosis | All diagnosis data is collected in a time-stamped fashion between January 2015 and December 2019; diagnosis is reported within the year, but not in a specific month/day
  Self-reported diagnosis of chlamydia
Gonorrhea diagnosis | All diagnosis data is collected in a time-stamped fashion between January 2015 and December 2019; diagnosis is reported within the year, but not in a specific month/day
  Self-reported diagnosis of gonorrhea
Sexually transmitted diseases | All diagnosis data is collected in a time-stamped fashion between January 2015 and December 2019; diagnosis is reported within the year, but not in a specific month/day
  Self-reported diagnosis of any STD
Percent of time that condoms were used in sexual intercourse | 12 months
  Self-reported condom adherence
Number of ongoing sexual relationships | Through study completion, approximately 2 months
  Self-reported number of concurrent sexual partners
Number of sexual partners over the past 12 months | 12 months
  Self-reported number of sexual partners over the past 12 months
Selecting a potential date with many recent partners | Through study completion, approximately 2 months
  The likelihood of selecting a potential date with 6 or more recent sexual partners in the conjoint experiment. Both AMCEs (average marginal component effects) and marginal means will be computed, see statistical analysis plan.
  As part of a conjoint experiment the investigators expose participants to a partner selection task.
  The attributes in the experiment and possible attribute values can be seen below:
  Race/ethnicity: White/Black/Asian Education: High school/Undergraduate degree/Graduate degree Number of sexual partners (past 3 months): 1/2-5 partners/6 or more Recreational drug use: Never/Sometimes/Often Seeking a...: Committed relationship/Casual relationship Use of condoms: Occasional/Frequent
Selecting a potential date with frequent recreational drug use | Through study completion, approximately 2 months
  The likelihood of selecting a potential date with frequent recreational drug use in the conjoint experiment. Both AMCEs (average marginal component effects) and marginal means will be computed, see statistical analysis plan.
  As part of a conjoint experiment the investigators expose participants to a partner selection task.
  The attributes in the experiment and possible attribute values can be seen below:
  Race/ethnicity: White/Black/Asian Education: High school/Undergraduate degree/Graduate degree Number of sexual partners (past 3 months): 1/2-5 partners/6 or more Recreational drug use: Never/Sometimes/Often Seeking a...: Committed relationship/Casual relationship Use of condoms: Occasional/Frequent
Selecting a potential date with occasional condom adherence | Through study completion, approximately 2 months
  The likelihood of selecting a potential date with occasional condom use in the conjoint experiment. Both AMCEs (average marginal component effects) and marginal means will be computed, see statistical analysis plan.
  As part of a conjoint experiment the investigators expose participants to a partner selection task.
  The attributes in the experiment and possible attribute values can be seen below:
  Race/ethnicity: White/Black/Asian Education: High school/Undergraduate degree/Graduate degree Number of sexual partners (past 3 months): 1/2-5 partners/6 or more Recreational drug use: Never/Sometimes/Often Seeking a...: Committed relationship/Casual relationship Use of condoms: Occasional/Frequent

OTHER OUTCOMES:
The likelihood at which a respondent would engage a partner in casual sex with without using condoms | Through study completion, approximately 2 months
  This is collected as a follow-up question for each profile in the conjoint experiment as detailed above

CONTACTS AND LOCATIONS:
Overall Officials: Kinga R Makovi, PhD, Principal Investigator — New York University Abu Dhabi
Locations (1):
- New York University Abu Dhabi, Abu Dhabi, United Arab Emirates